CLINICAL TRIAL: NCT05923047
Title: Mepolizumab and In-office Nasal Polypectomy in Patients With Chronic Rhinosinusitis (CRS). A Three Arm Study.
Acronym: MELYSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDIVAL
Record Dates: First submitted 2023-06-01; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Rhinosinusitis Chronic; Polyp, Nasal
MeSH Terms: conditions — Nasal Polyps | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: This trial includes three treatment arms.
  1. Combined group (In-office nasal polypectomy group with mepolizumab): This group will undergone in-office nasal polypectomy and will receive Mepolizumab.
  2. Medical group (mepolizumab): This group will receive Mepolizumab.
  3. Surgical group (In-office nasal polypectomy): This group will undergone in-office nasal polypectomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined group (Experimental): In-office nasal polypectomy group with mepolizumab
  Interventions: Drug: Mepolizumab
- Medical group (Experimental): (mepolizumab)
  Interventions: Drug: Mepolizumab
- Surgical group (Active Comparator): In-office nasal polypectomy
  Interventions: Procedure: Polypeptomy

INTERVENTIONS:
Drug: Mepolizumab — Patients in the Mepolizumab arms will receive 100 mg of subcutaneous mepolizumab every 4 weeks for a total of 12 doses in addition to daily topical corticosteroid treatment
  Arms: Combined group; Medical group
Procedure: Polypeptomy — This group will undergone in-office nasal polypectomy.
  Arms: Surgical group

SUMMARY:
This randomized, controlled multicenter trial will recruit patients aged 18 to 70 7 years with recurrent nasal polyposis requiring surgery and indication for biologic treatment according to EPOS 2020 guideline. Patients in the Mepolizumab arms will receive 100 mg of subcutaneous mepolizumab every 4 weeks for a total of 12 doses in addition to daily topical corticosteroid treatment.

All study procedures will be performed in five study visits and may take approximately 30 minutes. Clinical assessments include different questionnaires and nasal endoscopy. This trial includes three treatment arms.

1. Combined group (In-office nasal polypectomy group with mepolizumab): This group will undergone in-office nasal polypectomy and will receive Mepolizumab.
2. Medical group (mepolizumab): This group will receive Mepolizumab.
3. Surgical group (In-office nasal polypectomy): This group will undergone in-office nasal polypectomy. The main advantage is that it allows comparison of mepolizumab versus surgery and surgery/mepolizumab versus surgery + mepolizumab, providing more information on the most effective therapeutic approach.

The presence of adverse effects will be assessed in each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Participant 18 years of age or older
* Patients with a diagnosis of CRS with polyposis according to the criteria of the EPOS2020 guideline:

Chronic rhinosinusitis with nasal polyps in adults is defined as presence of two or more symptoms, one of which should be either nasal blockage / obstruction / congestion or nasal discharge (anterior / posterior nasal drip); ± facial pain/pressure; ± reduction or loss of smell; for ≥12 weeks; and either endoscopic signs of nasal polyps, and/or CT changes: mucosal changes within the ostiomeatal complex and/or sinuses.

* Patients with indication for biologic treatment according to the criteria of the EPOS2020 guideline. Presence of bilateral polyps in a patient who had ESS (except in cases where the patient is not fit for surgery, see bellow) and three of the following criteria are required:
* Evidence of type 2 inflammation (tissue eos> 10/hpf* or blood eos>250, OR total IgE> 100).
* Need for systemic corticosteroids or contraindication to systemic steroids (≥ 2 courses per yr, OR long term (>3 months)
* Significantly impaired quality of life (SNOT ≥ 40)
* Significant loss of smell (≥7 VAS)
* Diagnosis of comorbid asthma
* Basal eosinophil count (BEC) ≥300 cells/μL for surgical naïve patients- only those not fit for surgery (major criteria) or for those who have had surgery and have recurrence (minor criteria).
* Patients have been informed and signed consent to participate in the study.
* For those patients not suitable for surgery, the criteria of the EUFOREA guidelines for indication of biological treatment will be used (4 criteria, one of them being ≥300 cells/μL BEC).

Exclusion Criteria:

* Any serious or uncontrolled systemic or psychiatric illness that prevents a correct cognitive or endoscopic assessment or does not advise participation in the study.
* Unilateral localized secondary CRS (odontogenic, fungal ball, tumor).
* Bilateral diffuse secondary CRS (cystic fibrosis; eosinophilic granulomatosis with polyangiitis-S. de Churg-Strauss-; granulomatosis with polyangiitis-S de Wegener-; primary ciliary dyskinesia; selective immunodeficiencies.
* Pregnancy/ breast feeding
* Hypersensitivity to mepolizumab or it's excipients
* Patients unable to complete the questionnaire or follow prescribed treatment.
* Patients who are participating in another clinical trial related to polyposis or asthma.
* Previously documented failure with IL-5/IL-5 receptor biologics

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Mepolizumab+polypectomy compared to mepolizumab or polypectomy, using the change from baseline in sinonasal outcome test (SNOT-22) total score | up to 52 weeks

SECONDARY OUTCOMES:
Change in nasal polyposis severity VAS score at 4 weeks, 6 months, 12 months | up to 52 weeks
Change in endoscopic nasal polyp score at 4 weeks, 6 months, 12 months | up to 52 weeks
Improvement in individual VAS symptoms (rhinorrhea, mucus in throat, nasal blockage, and sense of smell), patient-reported outcomes at 4 weeks, 6 months, 12 months | up to 52 weeks
Number of patients no longer requiring rescue systemic corticosteroid treatment throughout the first year after the first month of starting the study | up to 52 weeks
Number of participants with mepolizumab and in-office nasal polypectomy related adverse events | up to 52 weeks
Change from baseline in sinonasal outcome test | up to 4 and 24 week
  The minimum value is 0 and maximum value is 110

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital de Curces, Bilbao
  - Hospital de Jerez, Jerez de la Frontera
  - Hospital Puerta del Hierro, Madrid
  - HUCA, Oviedo
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Virgen Macarena, Seville
  - Hospital Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: Undecided